CLINICAL TRIAL: NCT04917211
Title: Use of a Virtual Reality Mask in the Reduction of Pain and Anxiety During in Utero Surgical Procedures
Brief Title: Virtual Reality Mask During in Utero Surgical Procedures
Acronym: VIRTUALFETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP201134
Record Dates: First submitted 2021-04-29; First posted 2021-06-08 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Fetofetal Transfusion; Analgesia
Keywords: feotoscopy; virtual reality; fetal sugery
MeSH Terms: conditions — Fetofetal Transfusion; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual reality mask (Experimental): During the prior anesthesia consultation, the patient is informed of the possibility within the framework of the study of benefiting from analgesia with disconnection by a virtual reality mask, associated with local anesthesia. The patient will be explained that in the event of pain despite the virtual reality mask and local anesthesia, administration of remifentanil will be possible
  Interventions: Procedure: Virtual reality mask

INTERVENTIONS:
Procedure: Virtual reality mask — "The virtual reality mask is a mask with a screen that is put on the patient's face in the theatre before the surgery. It offers 3D scenarios of about 20 to 40 minutes on five different themes (the Zen garden, the mountain, the forest, the beach, the scuba diving) with music. The video-headset, equipped with head movement sensors, allows the 3D vision of a natural virtual world and the audio-headset emits sounds adapted to the virtual world and music therapy. The RV mask, via multi-sensorial immersion, focuses on two therapeutic targets which are pain and anxiety. It is a non-drug approach ""cousin"" to hypnosis. Its therapeutic effects are based on a distractive effect: attentive capture, an emotional effect: playfulness and positive suggestion, and a behavioral effect: the patient participates and is an actor in his care.
  "

SUMMARY:
"The virtual reality mask is an innovative technique, alternative to pharmacological medicine that would allow, in addition to its action on pain, to reduce anxiety and thus increase patient satisfaction by improving their experience of a risky situation. The therapeutic effects of the virtual reality mask are based on a distractive effect with attentive capture, an emotional effect due to ludic aspect and positive suggestion, and a behavioral effect.

In utero fetoscopy is a potentially painful procedure, particularly at the beginning of the procedure due to the introduction of a fetoscopy trocar in the amniotic cavity through the patient's uterus. It also generates anxiety in mothers because of the risks associated with the pathology and the procedure. This research focuses on the use of a virtual reality mask in the reduction of pain and anxiety during in utero surgical procedures.

The study is presented and proposed to the patient during the expert ultrasound examination by the obstetrician-gynecologist. Then the modalities are detailed by the anesthetist during the anesthesia consultation before the surgery. The patient is included in the study after the consent is signed. During the anesthesia consultation, the patient is informed of the possibility of analgesia through a virtual reality mask, associated with local anesthesia. It is explained that in case of pain despite the virtual reality mask and local anesthesia, remifentanil administration remains possible. During the anesthesia consultation, the patient's initial state of anxiety is assessed by the score Amsterdam Preoperative Anxiety and Information Scale.

The procedure takes place in the theatre room. Upon arrival in the theatre room (preoperative), an evaluation of the anxiety level is performed using a visual analog scale. The virtual reality mask is applied by the anesthesia team before skin disinfection and the placement of sterile drapes. During the procedure, a local anesthesia (non-adrenaline Xylocaine 1%) is performed as usual in order to insert the trocar in the amniotic cavity (diameter 3.5mm) which will be used to introduce the intra-amniotic fetoscope. If during the procedure, the patient feels pain, agitation, pain-related discomfort, morphine analgesia (Intravenous Remifentanil which means Intravenous Anesthesia with Objective Concentration) may be administered by the anesthesia team. Immediately after the procedure, the virtual reality mask will be removed.

DETAILED DESCRIPTION:
"The use of the virtual reality mask associated with local anesthesia during in utero fetal surgery procedures by fetoscopy in the treatment of complications of monochorionic twin pregnancies, could be an alternative to the use of intravenous remifentanil associated with local anesthesia. It would allow analgesia and reduction of patient anxiety, thus simplifying the procedure for both patients and surgeons.

The virtual reality mask is an innovative technique, alternative to pharmacological medicine that would allow, in addition to its action on pain, to reduce anxiety and thus increase patient satisfaction by improving their experience of a risky situation. The therapeutic effects of the virtual reality mask are based on a distractive effect with attentive capture, an emotional effect due to ludic aspect and positive suggestion, and a behavioral effect. The virtual reality mask has almost never been studied in a pregnant population, particularly in the context of in utero procedures associated with risks of fetal loss that further increase anxiety.

In utero fetoscopy is a potentially painful procedure, particularly at the beginning of the procedure due to the introduction of a fetoscopy trocar in the amniotic cavity through the patient's uterus. It also generates anxiety in mothers because of the risks associated with the pathology and the procedure. This research focuses on the use of a virtual reality mask in the reduction of pain and anxiety during in utero surgical procedures.

This is a prospective cohort study including pregnant women who have a complicated monochorionic twin pregnancy with an indication for fetal surgery (laser photocoagulation fetoscopy or Selective Termination of Pregnancy). The objective is to evaluate the success rate of the virtual reality mask for analgesia during fetoscopy in case of monochorionic twin pregnancies complicated. The success of the virtual reality mask for analgesia is defined by the absence of pain expressed by the woman (no administration of morphine (remifentanil)). The primary outcome is the administration or not of remifentanil. The secondary objectives are to evaluate firstly the variation in maternal anxiety when using the virtual reality mask, secondly the pain during the intervention and thirdly the maternal satisfaction.

The study is presented and proposed to the patient during the expert ultrasound examination by the obstetrician-gynecologist. Then the modalities are detailed by the anesthetist during the anesthesia consultation before the surgery. The presentation of the study and the signature of the consent can be done within two weeks prior to the procedure. The patient is included in the study after the consent is signed. During the anesthesia consultation, the patient is informed of the possibility of analgesia through a virtual reality mask, associated with local anesthesia. It is explained that in case of pain despite the virtual reality mask and local anesthesia, remifentanil administration remains possible. During the anesthesia consultation, the patient's initial state of anxiety is assessed by the APAIS score (Amsterdam Preoperative Anxiety and Information Scale). This is a validated score for the evaluation of patients' anxiety prior to a procedure. A score higher than 10 out of 20 indicates a high level of anxiety and helps to identify the most anxious patients. This score will therefore allow to evaluate the initial anxiety state by identifying two groups of patients according to their initial anxiety level: high (score strictly greater than 10) and normal (score less than or equal to 10), but also the mean initial anxiety score.

The procedure takes place in the theatre room. Upon arrival in the theatre room (preoperative), an evaluation of the anxiety level is performed using a visual analog scale.

The virtual reality mask is applied by the anesthesia team before skin disinfection and the placement of sterile drapes. During the procedure, a local anesthesia (non-adrenaline Xylocaine 1%) is performed as usual in order to insert the trocar in the amniotic cavity (diameter 3.5mm) which will be used to introduce the intra-amniotic fetoscope. This is a painful procedure because of the insertion of the trocar that crosses the abdominal wall, the subcutaneous tissue and the myometrium. Therefore, this justifies subcutaneous anesthesia up to the uterine serosa. If during the procedure, the patient feels pain, agitation, pain-related discomfort, morphine analgesia (Intravenous Remifentanil in IVAOC mode which means Intravenous Anesthesia with Objective Concentration) may be administered by the anesthesia team. Immediately after the procedure, the virtual reality mask will be removed. An evaluation of anxiety is performed using visual analog scale for anxiety. Maternal anxiety is thus evaluated by a score before and immediately after the intervention (variation in anxiety between before and after the intervention) (0 being the absence of anxiety and 10 being extremely intense anxiety). Moreover, the overall pain is assessed using visual analog scale for pain. Maternal pain will also be quantified in 2 ways: by the total dose of remifentanil (in relation to the total duration of the procedure) if remifentanil is administered and by a visual analog scale graded from 0 to 10 at the end of the intervention (0 being the absence of pain and 10 being the maximum pain imaginable). Lastly, the side effects sought are: nausea, dizziness, headaches, visual disturbances, discomfort.

The day after the intervention, an evaluation of the experience of the intervention and of maternal satisfaction will be performed using an EVAN-LR questionnaire. The EVAN-LR questionnaire is a validated satisfaction questionnaire for patients who remained conscious during the procedure. One of the strengths of this scale is its applicability in current practice as only 19 items need to be completed by the patient. The average filling time of the EVAN-LR is five minutes. For each item, the patient may check one of the following boxes: Not at all/ A little bit/ Moderately/ A lot/ Very much. If this was not possible the day after the operation, it is possible to fill it up to the second day after the operation. Patient participation ends after filling out the satisfaction questionnaire on day 1 or at the latest on day 2 after intervention. Patients will then be managed according to the usual practice.

The success rate of the virtual reality mask expected according to our experience is around 95%. In order to meet the objective of estimating this success rate with a good precision, the number of patients to be recruited is 73 patients having used the mask. This allows a precision of ±5.0% if the percentage of success is 95%, which seems a quite acceptable precision. In order to have useful data for a future therapeutic trial where there will be controls, the same data as for the participating women will be recorded for the women who refused the mask. Between 10 and 15 women who refused the virtual reality mask are expected to participate."

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old
* Complicated biamniotic monochorionic twin pregnancy
* Indication for fetal surgery: Fetoscopy laser photocoagulation or Selective termination of pregnancy.
* Patient Consent
* Affiliation to a social security coverage

Exclusion Criteria:

* No understanding of the French language
* Visually impaired or hard of hearing
* Participation in another intervention research
* Patient under State medical aid
* Psychiatric disorders (schizophrenia, schizophreniform disorders)
* Major neurocognitive disorders (dementias)
* Migraine helped a basic treatment
* Epilepsy with treatment
* Pacemaker carrier
* With lesions on the scalp

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the orimary outcome is the success of the virtual reality mask for analgesia defined by the absence of pain expressed by the woman (no administration of morphine (remifentanil)). | 2 days after the end of intervention
  "administration of remifentanil: no=success; yes=failure".

SECONDARY OUTCOMES:
Maternal anxiety | Baseline and immediately after the intervention
  Anxiety will be assessed by a Visual Analog Scale before and immediately after the intervention (0 being no anxiety and 10 being extremely intense anxiety). An assessment of anxiety using a visual analog scale will be performed before the procedure on arrival in the theatre room and immediately after the procedure after removing the VR mask. This scale provides a score from 0 to 10 to measure the anxiety felt by the patient. This before-after anxiety assessment is used to study the variation in the patient's anxiety between the beginning of the procedure and the end of the procedure.
The total dose of remifentanil in microgram (in relation to the total duration of the intervention) in case of administration of remifentanil | 2 days after the end of intervention
Overall maternal satisfaction | The satisfaction questionnaire is filled out on day 1 or at the latest on day 2 after intervention
  Evaluation of the experience of the intervention and of maternal satisfaction will be performed using an EVAN-LR questionnaire. The EVAN-LR questionnaire is a validated satisfaction questionnaire for patients who remained conscious during the procedure. One of the strengths of this scale is its applicability in current practice as only 19 items need to be completed by the patient. The average filling time of the EVAN-LR is five minutes. For each item, the patient may check one of the following boxes: Not at all/ A little bit/ Moderately/ A lot/ Very much.
Side effects | 2 days after the end of intervention
  nausea, dizziness, headaches, visual disturbances, discomfort
The rate of patients with a chosen virtual reality theme | 2 days after the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hanane BOUCHGHOUL, Principal Investigator — Public Assistance of Paris Hospitals
Locations (1):
- Hannane BOUCHGHOUL, Le Kremlin-Bicêtre, France